CLINICAL TRIAL: NCT00035113
Title: An Open-Label Phase IIa Trial Evaluating the Safety and Efficacy of EPO906 as Therapy in Patients With Androgen-independent Prostate Cancer
Brief Title: EPO906 Therapy in Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2204
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Prostatic Neoplasms
Keywords: prostate cancer; prostate; androgen independent; cancer; tumor; tumour; neoplasm; carcinoma; intravenous; epothilone
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Carcinoma | interventions — epothilone B

INTERVENTIONS:
Drug: epothilone b

SUMMARY:
This study will examine whether the new investigational drug EPO906, given by intravenous infusion (IV directly into the vein), is effective in shrinking tumors and preventing the growth of cells that cause prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

The following patients may be eligible for this study:

* Patients with any histologically proven prostate cancer with measurable metastatic disease or PSA progression > 20ng/ml after initial hormonal therapy will be eligible
* Patients must be maintained on androgen ablation therapy with a LHRH agonist or have undergone orchiectomy
* Patients in whom bicalutamide or flutamide has been recently withdrawn must demonstrate progression of disease and be at least 6 weeks and 4 weeks respectively, beyond the discontinuation of such agents
* Patients taking PC-SPES must discontinue therapy for a minimum of 4 weeks
* For patients with disease progression defined solely by PSA increase: two consecutive rises in PSA measurement, over a 4-week period (each separated from the previous by 2 weeks) - the last measurement must be at least 50% greater than the nadir PSA achieved after the last therapeutic maneuver
* For patients who discontinued bicalutamide therapy prior to study entry, a third rising PSA measurement is required 2 weeks from the second PSA measurement (i.e. over a 6 week period)
* Must have a life expectancy of greater than three (3) months
* Bilirubin must be within normal limits. Transaminases (SGOT and/or SGPT) may be up to 2.5 X institutional upper limit of normal if alkaline phosphatase is less than the upper limit of normal, or alkaline phosphatase may be up to 4 X upper limit of normal if transaminases are less than or equal to the upper limit of normal
* For patients with disease progression defined by measurable disease: changes in measurable size of lymph nodes or parenchymal masses on physical or radiologic examination (bone scan findings are not adequate to assess measurable disease).

Exclusion Criteria:

The following patients are not eligible for the study:

* Patients with symptomatic CNS metastases or leptomeningeal involvement
* Patients with any peripheral neuropathy or unresolved diarrhea greater than Grade 1
* Patients with severe cardiac insufficiency
* Patients taking Coumadin or other warfarin-containing agents with the exception of low dose Coumadin (1 mg or less) for the maintenance of in-dwelling lines or ports
* Patients who received palliative radiotherapy to tumors located centrally less than 4 weeks (28 days) prior to planned enrollment date (palliative radiotherapy to isolated peripheral bone metastases is allowed)
* Patients experiencing hormone withdrawal syndrome, or are 28 days post-withdrawal of anti-androgen therapy (42 days for bicalutamide)
* Patients who have had more than one prior chemotherapy regimen for hormone-resistant metastatic disease
* Patients with disease measurable only by bone scan
* Patients who have received corticosteroids within the past 28 days (may be waived with approval from Novartis)
* History of another malignancy within 5 years prior to study entry except curatively treated non-melanoma skin cancer
* Patients who have undergone major surgery for any cause less than 4 weeks prior to study entry
* Patients with radiation therapy or chemotherapy within the last four weeks
* Patients with active or suspected acute or chronic uncontrolled infection including abcesses or fistulae
* HIV+ patients

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-01; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Tumor response as assessed by radiologic techniques and/or physical examination based on Response Evaluation Criteria in Solid Tumors (RECIST)

SECONDARY OUTCOMES:
Time to progression
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - Pacific Shores Medical Group, Long Beach, California
  - California Pacific Medical Center, San Francisco, California
  - University of Maryland - Greenbaum Cancer Center, Baltimore, Maryland
  - Cancer Institute of New Jersey (CINJ), New Brunswick, New Jersey
  - Seattle Cancer Care Alliance, Seattle, Washington